CLINICAL TRIAL: NCT01059266
Title: A Prospective, Randomized, Open, Multi-centre Study to Assess Safety of PURETHAL Grasses Given With a Rush Induction Schedule to Patients With Allergic Rhinoconjunctivitis
Brief Title: PURETHAL Grasses Rush Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HAL Allergy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P/0035
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Allergic Rhinitis; Allergic Rhinoconjunctivitis
Keywords: immunotherapy; grass pollen; seasonal allergy; dose tolerability
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional regimen of PURETHAL Grasses (Active Comparator): Initial treatment:
  6 incremental weekly subcutaneous doses of 0.05, 0.1, 0.2, 0.3, 0.4 and 0.5 ml (week 1, 2, 3, 4, 5, 6).
  Maintenance treatment:
  0.5 ml in intervals according to registered scheme (week 8, 10, 12, 16).
  Interventions: Drug: PURETHAL Grasses, 20.000 AUM/ml
- rush regimen of PURETHAL Grasses (Experimental): Initial treatment:
  3 incremental weekly subcutaneous doses of 0.1, 0.3, and 0.5 ml (week 1, 2, 3)
  Maintenance treatment:
  3 monthly doses of 0.5 ml (week 7, 11, 15).
  Interventions: Drug: PURETHAL Grasses, 20.000 AUM/ml

INTERVENTIONS:
Drug: PURETHAL Grasses, 20.000 AUM/ml — subcutaneous injections of increasing doses according to the described regimen

SUMMARY:
This study investigates the safety of two up-dosing regimen. The safety of PURETHAL Grasses will be evaluated in a rush regimen (maximum dose reached in 3 injections during 2 weeks) compared to the conventional regimen (maximum dose reached in 6 injections during 5 weeks).

The primary parameter will be the proportion of patients who experience systemic reactions > grade I within 24 hours after injection or who need more than 2 additional injections during the up-dosing phase until the maintenance dose has been reached.

It is expected that up-dosing PURETHAL Grasses according to the rush regimen is as safe as using the conventional regimen.

ELIGIBILITY:
Inclusion Criteria

* Patients with rhinitis or rhinoconjunctivitis, with or without mild asthma (FEV1 > 70%) for at least 2 years related to grass pollen, eligible for SCIT.
* Confirmation of IgE-mediated allergy by means of:

  * Positive SPT to grass pollen (mean wheal diameter ≥ 3 mm and negative control truly negative (no reaction), or
  * Specific serum IgE-test (ssIgE >0.7 U/ml) for grass pollen, or
  * Positive provocation test for grass pollen.
* Age ≥ 18 years.
* Patients have given a written informed consent

Exclusion Criteria:

* Chronic asthma or emphysema, particularly with a FEV1 ≤ 70% of predicted value.
* Serious immuno-pathological diseases or malignancies (including auto-immune diseases, tuberculosis, HIV).
* Active inflammation/infection of the target organs (nose, eyes, lungs).
* Severe atopic dermatitis in need for systemic immunosuppressive medication.
* Symptomatic coronary heart diseases (e.g heart failure, recent myocardial infarction, unstable angina, serious arrhythmias) or severe (even under treatment) arterial hypertension.
* Severe kidney disease.
* Diseases with a contra-indication for the use of adrenaline.
* Treatment with systemic or local beta-blockers or immunosuppressive drugs.
* History of life threatening anaphylactic events, including anaphylactic food allergy, insect venom anaphylaxis, exercise or drug induced anaphylaxis.
* Any specific immunotherapy (including sublingual) during the study period or during the previous 3 years for a period longer than three months.
* Participation in a clinical study with a new investigational drug within the last three months.
* Pregnancy, lactation or inadequate contraceptive measures (adequate measures: oral contraceptives, IUD, condom use if used together with a spermicide and having no sexual relationship with a man).
* Alcohol or drug abuse.
* Lack of co-operation or severe psychological disorders.
* Completed or ongoing long-term treatment with tranquilizer or psycho active drugs.
* Low compliance or inability to understand instructions/study documents.
* Completed or ongoing treatment with anti-IgE-antibody.
* Patients being in relationship or dependence with the sponsor or investigator.
* Allergy to any of the excipients.
* Severe illness or any other condition, which makes the patient, in the opinion of the investigator, unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-02; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
systemic reactions > grade I or large local reactions related to injection | 24 hrs after injection

SECONDARY OUTCOMES:
specific serum IgE and IgG concentrations | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Pfaar, MD, Study Chair — Zentrum für Rhinologie & Allergologie, An den Quellen 10, D - 65183 Wiesbaden
Locations (11):
- Germany (11):
  - Universitätsklinikum Bonn Klinik u. Poliklinik f. Dermatologie, Bonn
  - Practice Blum, Dortmund
  - Uni-Klinikum Carl Gustav Carus Klinik und Poliklinik für HNO, Dresden
  - Practice Thieme, Duisburg
  - Medaimun GmbH, Frankfurt
  - Practice Wrede, Herford
  - Dr. med. Jörg Michael Nebel, Koblenz
  - Practice Scholz, Mahlow
  - St. Kamillus Krankenhaus Abt. Lungen- und Bronchialheilkunde und Allergologie, Mönchengladbach
  - Practice Termeer, Stuttgart
  - Zentrum für Rhinologie & Allergologie, Wiesbaden